CLINICAL TRIAL: NCT02412514
Title: Assessing the Intestinal and Humoral Immunity of Sequential Schedules of Inactivated Poliovirus Vaccine and Bivalent Oral Poliovirus Vaccine for Routine Childhood Immunization in Bangladesh
Brief Title: Intestinal and Humoral Immunity of Sequential Polio Vaccination Schedules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-14114
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-04

CONDITIONS: Poliomyelitis
Keywords: polio; inactivated poliovirus vaccine; oral poliovirus vaccine; IPV; OPV
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Infants assigned to Arm A will receive bOPV at 6, 10, and 14 weeks of age and IPV at 6 weeks of age.
  Interventions: Biological: bOPV (three dose); Biological: IPV
- Arm B (Active Comparator): Infants assigned to Arm B will receive bOPV at 10 and 14 weeks of age and IPV at 6 weeks of age.
  Interventions: Biological: bOPV (two dose); Biological: IPV

INTERVENTIONS:
Biological: bOPV (three dose) — bOPV administered at 6, 10, and 14 weeks of age.
  Arms: Arm A
Biological: bOPV (two dose) — bOPV administered at 10 and 14 weeks of age.
  Arms: Arm B
Biological: IPV — IPV administered at 6 weeks of age

SUMMARY:
This is a phase IV open-label randomized clinical trial that will compare intestinal and humoral immunity in infants receiving inactivated poliovirus vaccine (IPV) and two or three doses of bivalent oral poliovirus vaccine (bOPV).

DETAILED DESCRIPTION:
The goal of polio vaccination is to protect the individual from paralytic disease (humoral immunity) and to prevent transmission of poliovirus (intestinal immunity). Inactivated poliovirus vaccine (IPV) induces humoral (systemic) immunity to all three types of poliovirus (1, 2 and 3), protecting individuals from developing paralytic polio when exposed to wild type poliovirus. However, it induces little intestinal immunity. Intestinal immunity inhibits poliovirus replication thereby reducing the quantity and duration of poliovirus excretion in stool. This is critical in preventing the spread of poliovirus to others.

Oral polio vaccines are live attenuated vaccines and trivalent OPV (tOPV) is a mixture of poliovirus strains type 1, 2 and 3. Like IPV, OPV induces humoral immunity and is more effective than IPV at inducing intestinal immunity. In most developing countries, routine childhood immunization for poliovirus consists of three doses of tOPV at 6, 10 and 14 weeks of age and may also include a birth dose of tOPV.

An important limitation is that the vaccine virus in OPV can mutate and acquire neurovirulence causing paralysis either due to vaccine-associated paralytic polio (VAPP) or due to circulating vaccine-derived polioviruses (cVDPVs), in which the attenuated vaccine virus not only acquires the ability to cause paralysis but can also circulate similarly to wild poliovirus (WPV). The potential of vaccine virus to acquire neurovirulence and cause paralytic poliomyelitis is incompatible with eradication of polio. Therefore, polio eradication will require eventual cessation of all OPVs.

The last case of WPV type 2 was reported in 1999 in India. Type 2 vaccine virus in tOPV is most likely to cause cVDPVs and over 80% of cVDPVs over the past decade have been cVDPV2. Of the estimated 250-500 annual VAPP cases, almost 40% are due to type 2. Thus, with the eradication of WPV2 it is imperative to prioritize removal of type 2 containing OPV.

The licensing and availability of bOPV containing type 1 and 3 offers the option of an OPV that does not contain OPV2. In April 2013, the Strategic Advisory Group of Experts on Immunization (SAGE) recommended phased cessation of OPVs starting with the switch from tOPV to bOPV. After the switch, bOPV is expected to be administered at 6, 10 and 14 weeks of age, the typical routine poliovirus immunization schedule in developing countries for tOPV. Additionally, at least one dose of IPV was recommended to prevent rapid rise in type 2 susceptibility in the birth cohorts born after the switch to bOPV.

The Global Polio Eradication Initiative (GPEI) has advocated for administration of at least one dose of IPV and delaying the dose to 14 weeks of age to decrease interference by maternal antibodies and provide the highest seroconversion possible with a single dose of IPV in the Expanded Program on Immunization (EPI) schedule. The GPEI position of introducing only one dose of IPV at 14 weeks of age is principally based on findings from a trial in Cuba that reported type 2 seroconversion of 63% with a single dose of IPV given at 16 weeks of age. The current schedule of Bangladesh is tOPV at 6, 10 and 14 weeks of age with IPV also at 14 weeks of age.

As a result of the addition of IPV to the routine immunization schedule, children will receive four doses of the polio vaccine (three bOPV and one IPV) but are four doses necessary? Could IPV administered with a reduced number of bOPV doses still lead to protective levels of humoral and intestinal immunity? Previous studies in the US and UK suggest that two doses of OPV given with one or two doses of IPV induces protective levels of humoral and intestinal immunity comparable to three doses of tOPV. Furthermore, a recent study in Bangladesh found that there were no significant differences in type 1 or 3 seroconversion proportions among children on a three-dose bOPV schedule versus a fractional IPV (f-IPV)/bOPV schedule (two f-IPV, one bOPV). Although there were significant differences in vaccine virus excretion among children who received only bOPV compared to f-IPV/bOPV to type 1 and 3, this difference could have been diminished if a second dose of bOPV was given instead of f-IPV .

In addition, there has been interest in whether a VAPP-protective schedule could mount protective levels of immunity in individuals. A VAPP-protective schedule is the administration of IPV as the first dose of poliovirus vaccination. The risk of VAPP is highest with the first dose of OPV and diminishes with subsequent OPV administrations. There is no risk of VAPP when IPV is given as the first dose because the vaccine uses killed virus. The rationale behind the VAPP-protective schedule is that individuals would have prior exposure to types 1, 2, and 3 through IPV before their first bOPV administration, thereby decreasing the risk for VAPP.

Investigators of this trial will assess if a reduced number of bOPV doses given with a dose of IPV confers a protective level of immunity against polio by examining the intestinal and humoral immunity induced by two different bOPV/IPV VAPP-protective sequential schedules among infants in Bangladesh. Specially, investigators will examine the proportion of seroconversion and vaccine virus excretion in children who receive an IPV dose at 6 weeks of age and bOPV at 6, 10 and 14 weeks of age in comparison to children who receive an IPV dose at 6 weeks of age and bOPV only at 10 and 14 weeks of age.

Setting: Mirpur is a suburb of Dhaka with a population of about one million in an area of 59 square kilometers. Mirpur Thana of Dhaka city is divided into 14 sections. Mirpur is about 8 kilometers from icddr,b's Dhaka Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute diarrhea, infection or illness at the time of enrollment (6 weeks of age) that would require infant's admission to a hospital or would contraindicate provision of OPV per country guidelines.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age).
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine or contents of polio vaccine.
* Infants from multiple births. Infants from multiple births will be excluded to reduce the potential for contact transmission of vaccine poliovirus to siblings. The infant(s) from a multiple birth who is/are not enrolled would be likely to receive routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).

Ages: 6 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 456 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in type 1 and 3 excretion of vaccine poliovirus particles in stool one week after administration of the bOPV challenge dose. | One week
Change in type 1, 2 and 3 poliovirus antibody responses prior to administration of poliovirus vaccinations compared to after completion of poliovirus vaccinations. | 12 weeks

SECONDARY OUTCOMES:
Change in type 1 and 3 excretion of vaccine poliovirus in stool two weeks after administration of the bOPV challenge dose at 18 weeks of age. | Two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mirpur Clinic (International Centre for Diarrhoeal Disease Research, Bangladesh), Dhaka, Bangladesh

REFERENCES:
- [Derived] Snider CJ, Zaman K, Estivariz CF, Aziz AB, Yunus M, Haque W, Hendley WS, Weldon WC, Oberste MS, Pallansch MA, Wassilak SGF, Anand A. Assessing the mucosal intestinal and systemic humoral immunity of sequential schedules of inactivated poliovirus vaccine and bivalent oral poliovirus vaccine for essential immunization in Bangladesh: An open-label, randomized controlled trial. Vaccine. 2024 Sep 17;42(22):126216. doi: 10.1016/j.vaccine.2024.126216. Epub 2024 Aug 14. PMID 39146859